CLINICAL TRIAL: NCT05736991
Title: Deep Learning Signature Based on PET-CT Images for Predicting the Novel Grading System of Clinical Stage I Lung Adenocarcinoma
Brief Title: Deep Learning Signature for Predicting the Novel Grading System of Clinical Stage I Lung Adenocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: Ningbo No.2 Hospital (Other); Zunyi Medical College (Other); The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Chang Chen, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: DLGS
Record Dates: First submitted 2023-02-07; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Lung Adenocarcinoma; Radiomics; Grading System
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PET/CT-based Radiomics Signature — Radiomics Signature Based on PET-CT for Predicting the Novel Grading System of Clinical Stage I Lung Adenocarcinoma

SUMMARY:
The purpose of this study is to evaluate the performance of a PET/ CT-based deep learning signature for predicting the grade 3 tumors based on the novel grading system in clinical stage stage I lung adenocarcinoma based on a multicenter prospective cohort.

ELIGIBILITY:
Inclusion Criteria:

(1) Participants scheduled for surgery for radiological finding of pulmonary lesions from the preoperative thin-section CT scans; (2) The maximum diameter of lesion less than 4 cm on CT scans; (3) The maximum short axis diameter of lymph nodes less than 1 cm on CT scan; (4) The SUVmax of hilar and mediastinal lymph nodes less than 2.5; (5) Pathological confirmation of primary lung adenocarcinoma; (5) Age ranging from 20-75 years; (6) Obtained written informed consent.

Exclusion Criteria:

(1) Multiple lung lesions; (2) Poor quality of PET-CT images; (3) Participants with incomplete clinical information; (4) Mucinous adenocarcinomas; (5) Participants who have received neoadjuvant therapy.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinical Stage I Lung Adenocarcinoma
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic curve | 2022.11-2023.4
  Area under the receiver operating characteristic curve

SECONDARY OUTCOMES:
Sensitivity | 2022.11-2023.4
  Sensitivity
Specificity | 2022.11-2023.4
  Specificity
Positive predictive value | 2022.11-2023.4
  Positive predictive value
Negative predictive value | 2022.11-2023.4
  Negative predictive value
Accuracy | 2022.11-2023.4
  Accuracy

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shanghai Pulmonary Hospital, Yangpu, Shanghai Municipality
  - Ningbo HwaMei Hospital, Ningbo, Zhejiang